CLINICAL TRIAL: NCT05078268
Title: Effect of HRV Biofeedback as Adjunctive Therapy to Self-help Cognitive Behavioral Therapy on Insomnia: A Pilot Randomized Controlled Trial
Brief Title: Heart Rate Variability Biofeedback as Adjunctive Therapy to Self-help CBT-I
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSY016
Record Dates: First submitted 2021-10-04; First posted 2021-10-14 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Insomnia
Keywords: HRV biofeedback; Self-help CBT-I; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined group (Experimental): Participants in combined group will receive both HRV biofeedback training and self-help CBT-I concurrently.
  Interventions: Behavioral: HRV biofeedback training and self-help CBT-I
- Self-help CBT-I only group (Active Comparator): Participants in self-help CBT-I only group will receive self-help CBT-I only.
  Interventions: Behavioral: Self-help CBT-I only

INTERVENTIONS:
Behavioral: HRV biofeedback training and self-help CBT-I — Participants will receive a booklet with content related to both self-help CBT-I and HRV biofeedback per week for 6 consecutive weeks. Participants are required to use around 1 hour to read through the content and perform the HRV biofeedback practice for around 20 minutes a day, 5-7 days a week and record their practice.
  Arms: Combined group
Behavioral: Self-help CBT-I only — Participants will receive a booklet with content related to self-help CBT-I only per week for 6 consecutive weeks. Participants are required to use 30 to 40 minutes to read through the content.
  Arms: Self-help CBT-I only group

SUMMARY:
This study will examine the effect of Heart Rate Variability (HRV) biofeedback as adjunctive therapy to self-help Cognitive Behavioral Therapy on insomnia (CBT-I) in Chinese adult population. Heart Rate Variability Biofeedback is a therapy training aiming at increasing heart rate oscillations through real-time feedback and slow breathing training. Several literature has found that HRV biofeedback training is effective in improving HRV and improving sleep quality and sleep efficiency (Gevirtz, 2013; Lin et al., 2019). On the other hand, self-help CBT-I is well-studied in efficacy of improving cognition and behaviors and relieving insomnia (Ho et al., 2014). Rare research study HRV biofeedback as adjunctive therapy to self-help CBT-I (Lehrer, 2017). In the light of this, this study will compare the efficacy of combination of both treatments with that of CBT-I alone, examining whether HRV biofeedback's focus on psychophysiological domain can help self-help CBT-I in more significantly improving HRV and sleep quality.

DETAILED DESCRIPTION:
This study will be a pilot randomized controlled trial on the efficacy of HRV biofeedback as adjunctive therapy to self-help CBT-I on insomnia. Potential participants will be recruited from the community through posters, social media sites and/or emails. Prior to all study procedures, the research purpose and data collection procedure will be given to the participants and an informed consent will be obtained from potential participants. Around 44 eligible participants will be randomly assigned to either self-help CBT-I with HRV biofeedback (combined group) or self-help CBT-I only group in a ratio of 1:1. The randomization will be performed by an independent assessor using a computer-generated list of numbers. No deception is necessary. Participants in combined group will receive a booklet with content related to both self-help CBT-I and HRV biofeedback based on guidelines of self-help CBT-I and protocol for HRV biofeedback training per week for 6 consecutive weeks. Participants are required to use around 1 hour to read through the content. The combined group is requested to perform the HRV biofeedback practice with a Bluetooth sensor connected with Inner Balance mobile application for around 20 minutes a day, 5-7 days a week and record their practice. Self-help CBT-I only group will receive a booklet with content related to self-help CBT-I only per week for 6 consecutive weeks. Participants are required to use 30 to 40 minutes to read through the content. The combined group and self-help CBT-I only group will complete a set of questionnaires and HRV measurement before the treatment commences, immediately after treatment, and 4 weeks after the treatment sessions are completed.

ELIGIBILITY:
Inclusion Criteria:

1. Hong Kong residents aged 18-59 years
2. Cantonese language fluency
3. A global Insomnia Severity Index (ISI) score of 10 or higher [A cutoff score of 10 was optimal (86.1% sensitivity and 87.7% specificity) for detecting insomnia cases (Morin, Belleville, Bélanger & Ivers, 2011)]
4. A willingness to provide informed consent and comply with the trial protocol

Exclusion Criteria:

1. have major psychiatric, medical or neurocognitive disorders that make participation infeasible or interfere with the adherence to intervention
2. previous suicide attempt, severe active suicidal ideation with a specific plan, severe self-harm, active substance abuse, or a history of psychosis.
3. having cardiovascular diseases that affect the measure of heart rate variability
4. having severe lung infections, central respiratory failure, electrolyte imbalance, fever and other diseases affecting the heart activity
5. having with other organic diseases, previous history of arrhythmias (atrial fibrillation and frequent premature beats), hyperthyroidism, history of syncope and autonomic nervous system dysfunction
6. have insomnia due to specific medical conditions, side effects of medication intake or other sleep disorders
7. change in medication or its dosage 2 weeks before the baseline measurement

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-11-20 (Estimated); Primary Completion 2022-05-20 (Estimated); Study Completion 2022-07-20 (Estimated)

PRIMARY OUTCOMES:
Change in Heart Rate Variability - Inner Balance | Baseline, immediate post-treatment, and 4-week follow-up
  Participants will be instructed to wear an Inner Balance bluetooth sensor connected with a mobile application Inner Balance to practice HRV biofeedback for around 30 minutes a day, 5-7 days a week.
Change in Insomnia Severity Index (ISI) | Baseline, immediate post-treatment, and 4-week follow-up
  ISI is a 7-item scale designed to evaluate perceived insomnia severity. Ratings on the 5-point Likert scale are obtained on the perceived severity of sleep-onset, sleep-maintenance, early morning awakening problems, satisfaction with current sleep pattern, interference with daily functioning, noticeably of impairment attributed to the sleep problem, and level of distress caused by the sleep problem.
Change in Pittsburgh Sleep Quality Index (PSQI) | Baseline, immediate post-treatment, and 4-week follow-up
  The PSQI is a widely used 24-item scale used to access the sleep quality and disturbances over a 1-month interval. The 19 self-rated questions will be used, which is calculated by a seven-component score from: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping medication, and daytime dysfunction.

SECONDARY OUTCOMES:
Change in Pre-Sleep Arousal Scale (PSAS) | Baseline, immediate post-treatment, and 4-week follow-up
  The Pre-Sleep Arousal Scale (PSAS) includes 16 items scored on a 4-point Likert scale to assess pre-sleep arousal. PSAS includes two sub-scales: physical and cognitive arousals.
Change in Depression Anxiety Stress Scales (DASS-21) | Baseline, immediate post-treatment, and 4-week follow-up
  DASS-21 is a 21-items scales, comprises of three sub-scales which measures the negative emotional states of depression, anxiety, and stress, over the past week.
Change in The Multidimensional Assessment of Interoceptive Awareness, Version 2 (MAIA-2) | Baseline, immediate post-treatment, and 4-week follow-up
  The Multidimensional Assessment of Interoceptive Awareness (MAIA) is an 8-scale state-trait questionnaire with 37 items to measure multiple dimensions of interoception by self-report: Noticing, Not-Distracting, Not-Worrying, Attention Regulation, Emotional Awareness, Self-Regulation, Body Listening, and Trust.
Change in Sleep Locus of Control Scale (SLOC) | Baseline, immediate post-treatment, and 4-week follow-up
  The Sleep Locus of Control Scale (SLOC) is an 8-item questionnaire designed to evaluate a respondent's sleep-related locus of control - the degree to which an individual attributes his or her experiences of sleep to chance or to internal, intentional causes.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong